CLINICAL TRIAL: NCT01077336
Title: Clinical Outcomes in Candidemia Patients Based on in Vitro Susceptibility
Status: Completed | Type: Observational
Sponsor: University of Houston (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kevin W. Garey, Professor and Chair, University of Houston
Other Study IDs: G098881
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Blood Stream Infections; Candida
Keywords: susceptibility testing
MeSH Terms: conditions — Torulopsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized patients with candidemia

SUMMARY:
Susceptibility testing is commonly employed in patients with bacterial infections in order to guide rational use of antibiotics; however, the use of antifungal susceptibility testing is limited due to lack of availability, costs, and delays in receiving results. The goals of antifungal susceptibility testing should mirror those of antibacterial susceptibility testing: to predict clinical response or failure. Additionally, susceptibility reports should be used as a guide for physicians when transitioning patients from parenteral to oral antifungal agents. Currently, it is unknown whether antifungal susceptibility testing impacts treatment decisions in hospitals that routinely perform Candida susceptibility testing. The purpose of this study is to evaluate the changes in antifungal treatment based on in vitro susceptibility reports and how these decisions affect mortality, recurrence of infection, and length of hospital stay in candidemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with bloodstream infections due to Candida species

Exclusion Criteria:

* Patients will be excluded from this study if their medical charts contain incomplete outcome or susceptibility data. Patients treated empirically or definitively with amphotericin-based products will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a retrospective cohort study of 400 hospitalized patients with bloodstream infections from January 2006 to January 2009 due to Candida species
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Assess empiric choice of antifungal therapy in hospitalized patients with candidemia. | Assessments made for 30-days after postivie blood culture